CLINICAL TRIAL: NCT05752721
Title: Impact of Online Ordering on Low-Income Adults' Food Security in Online Food Pantry Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-01523
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Food Security

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Pantry Scheduled to Transition to Online Ordering (Experimental): Low-income adults who have visited the food pantry that is scheduled to transition to online ordering at least once. Participants will complete an in-person survey and a research assistant will record the food items they received in the relevant visit to the pantry. After the transition to online ordering at the intervention food pantry, participants will again complete the survey. Food selections for participants in the this arm will be accessible through the online ordering platform.
  Interventions: Behavioral: Transition to Online Ordering
- Food Pantry NOT Scheduled to Transition to Online Ordering (No Intervention): Low-income adults who have visited the food pantry that is NOT scheduled to transition to online ordering at least once. Participants will complete an in-person survey and a research assistant will record the food items they received in the relevant visit to the pantry. After the transition to online ordering at the intervention food pantry, participants will again complete the survey. Participants in this arm will record their food selections and send them to the study team.

INTERVENTIONS:
Behavioral: Transition to Online Ordering — The intervention food pantry will transition to online ordering at least once.
  Arms: Food Pantry Scheduled to Transition to Online Ordering

SUMMARY:
The primary objectives of this study are to determine whether the transition to online ordering at a choice-based food pantry network influences food security status among low-income adults and determining whether there are differences in impact by age group.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* have visited a food pantry that either is or is not scheduled to transition to online ordering at least once
* have capacity and willingness to provide consent
* speaks English

Exclusion Criteria:

* aged less than 18 years
* have not visited a food pantry that either is or is not scheduled to transition to online ordering at least once
* does not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Rummo, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research. After 36 months the data will be available in NYU Langone's data warehouse but without investigator support other than deposited metadata. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research. The informed consent form, clinical study report, and analytic code will also be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in NYU Langone's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Derived] Rummo P, Yi S, Seet C, Strahs L, Kong J, Jebejian D, Elbel B. The impact of online ordering on food security in a food pantry system in New York City. Transl Behav Med. 2025 Jan 16;15(1):ibaf031. doi: 10.1093/tbm/ibaf031. PMID 40539601

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Started | 114 | 90
Completed | 77 | 58
Not Completed | 37 | 32
Not completed — Lost to Follow-up | 22 | 20
Not completed — Withdrawal by Subject | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering | Total
Number analyzed (Participants) | 77 | 58 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (15.3) | 65.2 (17.2) | 59.1 (16.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 63 | 35 | 98
  Male | 9 | 23 | 32
  Other Gender | 2 | 0 | 2
  Unknown or not reported | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 61 | 44 | 105
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 8 | 6 | 14
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 7 | 16
  White | 49 | 40 | 89
  Middle Eastern or North African | 2 | 0 | 2
  More than one race | 3 | 1 | 4
  Unknown or not reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 77 | 58 | 135

OUTCOME MEASURES:

1. Primary Outcome: U.S. Household Food Security Survey Module: Six-Item Short Form Score
Description: 6-item assessment of food security. The total score ranges from 0-6, where: 5-6 = very low food security; 2-4 = low food security; and 0-1 = high or marginal food security.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 77 | 58
score on a scale | 3.6 (2.2) | 2.7 (2.3)

2. Primary Outcome: U.S. Household Food Security Survey Module: Six-Item Short Form Score
Description: as for outcome 1
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 77 | 58
score on a scale | 2.9 (2.3) | 2.0 (2.2)

3. Secondary Outcome: Time to Obtain Food From Food Pantry Per Visit
Description: Expressed in minutes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 114 | 90
minutes | 5.1 (11.1) | 27.7 (28.2)

4. Secondary Outcome: Time to Obtain Food From Food Pantry Per Visit
Description: Expressed in minutes.
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 77 | 58
minutes | 3.7 (4.3) | 29.4 (29.0)

5. Secondary Outcome: Composite Weekly Fruit & Vegetable Intake Score
Description: The Behavioral Risk Factor Surveillance System's 2017 six-item fruit and vegetable screener, where values correspond to the number of times a participant consumed fruits and vegetables per week as a composite score. The total score ranges from 0 to infinity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 114 | 90
score on a scale | 16.0 (12.4) | 18.1 (18.3)

6. Secondary Outcome: Composite Weekly Fruit & Vegetable Intake Score
Description: as for outcome 5
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 77 | 58
score on a scale | 16.1 (9.9) | 16.4 (7.6)

7. Secondary Outcome: Center for Nutrition & Health Impact's Household Nutrition Security Survey Module: Four-Item Short Form Score
Description: 4-item assessment of nutrition security. The four items within the measure are scored from 0 (if the participant selects "Always") to 4 (if the participant selects "Never"). The total score is the average of the four item scores and ranges from 0-4; higher scores indicate greater nutrition security, and scores of 2 or below indicate "low" levels of nutrition security.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 114 | 90
score on a scale | 3.6 (2.2) | 2.7 (2.3)

8. Secondary Outcome: Center for Nutrition & Health Impact's Household Nutrition Security Survey Module: Four-Item Short Form Score
Description: as for outcome 7
Time Frame: Month 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
Number analyzed (Participants) | 77 | 58
score on a scale | 2.9 (2.3) | 2.0 (2.2)

ADVERSE EVENTS:
Time Frame: 8 Month
Arm/Group | Food Pantry Scheduled to Transition to Online Ordering | Food Pantry NOT Scheduled to Transition to Online Ordering
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/90
Other Adverse Events (participants affected / at risk) | 0/114 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT05752721/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT05752721/ICF_000.pdf